CLINICAL TRIAL: NCT01602003
Title: A Multicenter, Multinational, Randomized, Active-controlled, Parallel Group, Double-blind, Phase III Trial to Evaluate the Efficacy and Safety of LC15-0444 Compared With Sitagliptin Added to Ongoing Metformin Therapy in Patients With Type 2 Diabetes Inadequately Controlled With Metformin Alone
Brief Title: Phase III Trial to Evaluate the Efficacy and Safety of LC15-0444 Compared With Sitagliptin Added to Ongoing Metformin Therapy in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-DPCL006
Record Dates: First submitted 2012-05-15; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444; BID protein, human; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- LC15-0444 25 mg bid (Experimental): LC15-0444 25 mg bid(twice daily)added on Metformin therapy
  Interventions: Drug: LC15-0444 25mg bid
- LC15-0444 50 mg qd (Experimental): LC15-0444 50 mg qd(once daily) added on Metformin therapy
  Interventions: Drug: LC15-0444 50mg qd
- Sitagliptin 100mg qd (Active Comparator): Sitagliptin 100 mg qd (once daily) added on the Metformin therapy
  Interventions: Drug: Sitagliptin 100mg qd

INTERVENTIONS:
Drug: LC15-0444 25mg bid — Each patient was given 3 different bottles of study drugs that comprised of two morning bottles and one evening bottles. Each morning bottle contained LC15-0444 25 mg or 50 mg or Sitagliptin 100mg(depending on the randomized group) or its matching placebo while the evening bottle contained LC15-0444 25 mg or its matching placebo. Patient was instructed to take 1 tablet from each bottle at regular times in the morning and evening every day during the 24-week double-blind treatment period.
  Arms: LC15-0444 25 mg bid
Drug: LC15-0444 50mg qd — Each patient was given 3 different bottles of study drugs that comprised of two morning bottles and one evening bottles. Each morning bottle contained LC15-0444 25 mg or 50 mg or Sitagliptin 100mg(depending on the randomized group) or its matching placebo while the evening bottle contained LC15-0444 25 mg or its matching placebo. Patient was instructed to take 1 tablet from each bottle at regular times in the morning and evening every day during the 24-week double-blind treatment period.
  Arms: LC15-0444 50 mg qd
Drug: Sitagliptin 100mg qd — Each patient was given 3 different bottles of study drugs that comprised of two morning bottles and one evening bottles. Each morning bottle contained LC15-0444 25 mg or 50 mg or Sitagliptin 100mg(depending on the randomized group) or its matching placebo while the evening bottle contained LC15-0444 25 mg or its matching placebo. Patient was instructed to take 1 tablet from each bottle at regular times in the morning and evening every day during the 24-week double-blind treatment period.
  Arms: Sitagliptin 100mg qd

SUMMARY:
Double-blind, randomized, multicenter, multinational (South Korea and India), parallel group study The study was divided into three parts: part 1 was a screening period started with an initial 2 weeks of exercise/diet program; part 2 was a double-blind treatment period during which eligible patients were randomized to Sitagliptin 100 mg qd (once daily), LC15-0444 25 mg bid (twice daily), or LC15-0444 50 mg qd groups and received the assigned treatment for 24 weeks; part 3 was for those patients who completed part 1 & 2 and consented to receive another 28 weeks of treatment with LC15-0444 50 mg qd.

Screening tests were performed on the patients who had given the written informed consent. After 2-week exercise/diet program according to the generally recognized guideline, eligible patients were assigned one of three treatment groups with 1:1:1 ratio. During the total of 24-week treatment period of part 2, each patient visited the study site at Week 6, 12, 18, and 24. Completing double-blind treatment for 24 weeks, each patient was asked to provide consent to participate in the part 3 of the study where all the patients were to receive LC15-0444 50 mg once daily. During 28-week treatment period of the part 3, each patient visited the study

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Type 2 Diabetes Mellitus
2. Adults between 18 and 75 years of age
3. Patients with HbA1c between 7% and 11%
4. Patients treated with metformin monotherapy for at least 12 weeks and treated with 1000 mg/day or higher dose of metformin for at least 4 weeks right before screening
5. Patients who signed on the consent form after informed on the object, method, and risks of the clinical study

Exclusion Criteria:

1. Patients with type 1 diabetes mellitus, gestational diabetes, or secondary diabetes
2. Patients who were taking or needed to take any drugs which may affect the control of blood glucose significantly (ex. glucocorticoids)
3. Patients who had experienced myocardial infarction, unstable angina or prior history of coronary artery bypass surgery within 6 months prior to screening, or patients with arrhythmia requiring treatment
4. Patients with NYHA class II-IV congestive heart failure
5. Patients with history of hepatic cirrhosis
6. Patients with renal failure or whose creatinine clearance was less than 60 ml/min
7. Patients with dysfunctional thyroid gland (with abnormal level of TSH)
8. Patients with ALT, AST or CPK exceeding 2.5 times of the upper limit of the normal range
9. Patients with BMI below 20 kg/m2 or exceeding 40 kg/m2
10. Patients with history of asthma or major skin allergy
11. Patients taking thyroid hormone, warfarin, dicoumarin or digoxin.
12. Patients with history of hypersensitivity to metformin or biguanides.
13. Patients with history of hypersensitivity to thiazolidinediones
14. Patients who took sodium channel blockers in the last 6 weeks prior to Visit 1.
15. Patients who were treated with insulin or glucagon-like peptide-1 (GLP-1) analogue or who took thiazolidinediones (Glitazone) in the last 6 months prior to Visit 1.
16. Patients with other reasons who the investigator decided not to be eligible for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change of HbAlc | from baseline to Week 24

SECONDARY OUTCOMES:
HbA1c Responder Rate | at Week 24
  responder rate of HbA1c <7%, <6.5% at week 24

CONTACTS AND LOCATIONS:
Overall Officials: Sun Woo Kim, MD, PhD, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- LG Life Sciences, Seoul, South Korea